CLINICAL TRIAL: NCT05720858
Title: The Effect of Aerobic Exercise Based Telerehabilitation Program on Upper Extremity Functıonality, Cognitive Status and Quality of Life in Patients With Survival Breast Cancer
Brief Title: Telerehabilitation in Survival Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Ramazan Cihad Yılmaz, lecturer, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/050
Record Dates: First submitted 2022-11-27; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Telerehabilitation; Exercise; Survival
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hospital group (Experimental): A total of 36 sessions (3 days a week) will be applied. Training intensity will be performed at the level of 4-6 according to the modified Borg scale, and rest will be allowed between exercises according to the tolerance of the patients. In the hospital-based group, a supervised aerobic exercise program will be applied in the hospital. There will be warm-up exercises before the exercise and cool-down exercises after. At the beginning of the session, warm-up exercises will begin. Flexibility exercises will be applied during the warm-up period. Warm-up and cool-down exercises will be performed for 10 minutes with 3 repetitions, including the upper and lower extremities and distal joints. Exercises will be performed for 3 months, with 10 repetitions in the first 6 weeks and 15 repetitions in the next 6 weeks.
  Interventions: Other: Aerobic exercise
- Telerehabilitation group (Experimental): A total of 36 sessions (3 days a week) will be applied. Training intensity will be performed at the level of 4-6 according to the modified Borg scale, and rest will be allowed between exercises according to the tolerance of the patients. Supervised sessions will be held with the telerehabilitation group via phone or computer video conference (For patients who agree to participate, the physiotherapist will initially conduct the first session face-to-face).
  There will be warm-up exercises before the exercise and cool-down exercises after. At the beginning of the session, warm-up exercises will begin. Flexibility exercises will be applied during the warm-up period. Warm-up and cool-down exercises will be performed for 10 minutes with 3 repetitions, including the upper and lower extremities and distal joints. Exercises will be performed for 3 months, with 10 repetitions in the first 6 weeks and 15 repetitions in the next 6 weeks.
  Interventions: Other: Aerobic exercise
- Control group (No Intervention): They will continue their routine activities. After the study, those who wish will be included in the exercise program.

INTERVENTIONS:
Other: Aerobic exercise — Reciprocal straight leg lift, Reciprocal hip knee flexion-extension, Lateral spinal rotation (Spinal rotation), Bridge Exercise, Elbow winging, Hip abduction, trunk extension, Shoulder elevation, Shoulder circulation, Shoulder flexion and extension, Shoulder abduction adduction, Reciprocal lateral trunk flexion and extension, Puching exercise, Mini Squat exercise, Reaching upward with hands reciprocally, Scapular adduction (Hands at waist), Push-ups on the wall, Knee Touch exercise, Arm Circles exercise, Reaching for feet in sitting position, Saw (The saw) exercise.
  Arms: Hospital group; Telerehabilitation group

SUMMARY:
The aim of this study is to determine the effect of telerehabilitation-based aerobic exercises on upper extremity functionality, cognitive status and quality of life in patients with survival breast cancer.

DETAILED DESCRIPTION:
Early detection of breast cancer and advances in treatment methods have led to an increase in survival after diagnosis. The prolongation of survival from breast cancer necessitated addressing the physical and psychosocial needs of individuals who have completed the active treatment process. Survival period breast cancer patients, need rehabilitation due to the delayed effects of treatment and difficulties encountered in everyday life. In the literature, the importance of exercise is emphasized in order to combat these problems. Physical activity levels are generally low in survival breast cancer patients, and many women reduce physical activity after diagnosis. Therefore, interventions are necessary to improve physical activity activity levels in breast cancer patients of the survival period.

In order to improve the physical activity levels of these patients, exercises can be performed in the hospital and at home. However, there may be problems in terms of adherence to exercise in interventions performed in the form of home exercise. That is why the importance of face-to-face, supervised exercises is reported in the literature. Supervised exercise can be offered in the hospital and in the form of telerehabilitation.

Telerehabilitation is considered as a promising alternative to conventional clinical rehabilitation programs by providing participation and transportation in health interventions. The simplest telerehabilitation system is used through video conferencing, in such a way that the therapist can monitor the patient remotely with the help of a camera. Telerehabilitation can be a valuable alternative education mode for patients who can manage technology at home but are unable or unwilling to participate in centre-based rehabilitation programs.

The aim of this study is to determine the effect of telerehabilitation-based aerobic exercises on upper extremity functionality, cognitive status and quality of life in patients with survival breast cancer.

Hypothesis 1: Aerobic-based telerehabilitation approach improves upper extremity functionality more than hospital-based exercise in surviving breast cancer patients.

Hypothesis 2: Aerobic-based telerehabilitation approach improves quality of life more than hospital-based exercise in surviving breast cancer patients.

Hypothesis 3: Aerobic-based telerehabilitation approach improves cognitive function more than hospital-based exercise in surviving breast cancer patients.

Exercises:

* Reciprocal straight leg lift
* Reciprocal hip knee flexion-extension
* Lateral spinal rotation (Spinal rotation)
* Bridge Exercise
* Elbow winging
* Hip abduction
* trunk extension
* Shoulder elevation
* Shoulder circulation
* Shoulder flexion and extension
* Shoulder abduction adduction
* Reciprocal lateral trunk flexion and extension
* Puching exercise
* Mini Squat exercise
* Reaching upward with hands reciprocally
* Scapular adduction (Hands at waist)
* Push-ups on the wall
* Knee Touch exercise
* Arm Circles exercise
* Reaching for feet in sitting position
* Saw (The saw) exercise

A total of 36 sessions (3 days a week) will be applied. Training intensity will be performed at the level of 4-6 according to the modified Borg scale, and rest will be allowed between exercises according to the tolerance of the patients. Supervised sessions will be held with the telerehabilitation group via phone or computer video conference (For patients who agree to participate, the physiotherapist will initially conduct the first session face-to-face). In the hospital-based group, a supervised aerobic exercise program will be applied in the hospital.

There will be warm-up exercises before the exercise and cool-down exercises after. At the beginning of the session, warm-up exercises will begin. Flexibility exercises will be applied during the warm-up period. Warm-up and cool-down exercises will be performed for 10 minutes with 3 repetitions, including the upper and lower extremities and distal joints.

Exercises will be performed for 3 months, with 10 repetitions in the first 6 weeks and 15 repetitions in the next 6 weeks. Evaluation will be done at baseline, 6 weeks, 12 weeks and 6 months. The exercises will be performed for 40 minutes for the first 6 weeks and 50 minutes for the next 6 weeks.

It is aimed to evaluate the effect of aerobic exercise-based telerehabilitation program on upper extremity functionality, cognitive status and quality of life in patients with survival breast cancer who meet the inclusion criteria. After signed informed consent, all participants will be randomized 1:1:1 to the telerehabilitation group, hospital-based exercise group, and control group using a computer-generated random number sequence. Computer generated random numbers (RESEARCH RANDOMIZER) will be used. Sample Size was determined using the G*Power system to suit power analysis procedures. Based on the power calculation EORTC QLQ-C30, the sample size of each group was determined as 19 with an effect size of 0.95 at 80% power (1). Considering possible patient losses, it was planned to recruit 20% more patients. In total, 69 patients of 23 patients are planned to be treated. The study is a mixed method type randomized controlled intervention study in which quantitative and qualitative research methods are used together. Sequential explanatory design: (QUANTITATIVE → qualitative) In this design, qualitative data is collected after predominantly quantitative data are collected and analyzed. Priority is usually in quantitative data. Qualitative data is mainly obtained to support quantitative data. Data analysis is interrelated and often combined in data interpretation and discussion sections. This design is particularly useful in explaining unexpected research findings or relationships. Questionnaires to be used during the evaluation;

* Patient Introductory Information Form
* Chronic Disease Treatment Functional Assessment Fatigue (FACIT Fatigue) Scale
* DASH (Arm, Shoulder and Hand Problems Questionnaire)
* The Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog)
* EORTC QLQ-C30 Quality of Life Scale

Qualitative questions to be used;

* What are the changes in upper extremity functionality after the treatment program?
* What are the changes have experienced in cognitive status after the treatment program?
* What changes have experienced in quality of life after the treatment program?
* What are the most important difficulties/gains have experienced in the post-treatment period?

After obtaining informed consent from the participants, they will be interviewed and asked about their experience using the telerehabilitation system and their intention to use the system in the future. Content analysis and inductive approach will be used in the evaluation of the data (Content analysis). In the analysis process, the in-depth interviews will be written down verbatim, the transcripts will be analyzed and the sections that form a meaningful whole in themselves will be named and coded by the researchers. Sub-themes that can bring together related codes will be determined. With the permission of the participants, their conversations will be audio recorded. Participants will be informed that they can stop the interview at any time. Afterwards, the data will be reported. In line with the themes investigators will reveal in the findings section, direct quotations of the participants about the research topic will be included (Patient names will be replaced with pseudonyms in order to protect the privacy of the participants). Expert support will be sought for qualitative data analysis (NVIVO qualitative software).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65
* Literate
* Having a diagnosis of breast cancer stage 1-2
* Complete breast cancer primary treatment at least 6 months before (excluding hormone therapy/aromatase inhibitors)
* Providing the cooperation
* Be woman
* Physically inactive (60 minutes of structured exercise per week <)
* Patients willing and voluntarily to participate in the study

Exclusion Criteria:

* Who are using one of the psychotic, anxiolytic, antidepressant, analgesic and sleeping pills
* With metastases
* Those with a history of lymphedema
* With neurological disease
* Those who are pregnant or breastfeeding
* Uncontrolled hypertensive patients
* Those incapable of verbal communication or physical movement
* Patients who did not agree to participate in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with survival period breast cancer will be taken
Enrollment: 69 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire) | A day before the treatment
  The EORTC-QLQ-C30 Quality of Life Scale includes 30 questions and three subheadings: general well-being, functional difficulties, and symptom control. The first 28 of the 30 items in the scale are a four-point Likert-type scale and the items are evaluated as Never: 1, A little: 2, Quite: 3 or A lot: 4 points. In the 29th question of the scale, the patient is asked to evaluate his health on a scale from 1 to 7 (1: Very poor and 7: Excellent), and in the 30th question, the general quality of life. The 29th and 30th questions constitute the general well-being area. High scores in this section indicate a high quality of life, and low scores indicate a decrease in quality of life. (Hospital group, telerehabilitation group and control group will be evaluated)
Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) | A day before the treatment
  This form evaluates the parameters of cognitive sensitivity (sharpness), attention and coordination, memory, verbal fluency, functional confusion, observations of others about the individual, change in functionality compared to before, and quality of life. It consists of 4 subtitles and 37 questions in total. Questions in the sections of perceived cognitive impairment, comments from other people, perceived cognitive skills, and impact on quality of life are scored between 0 and 4 (0-several times per day times, 4-never). In 9 questions in the field of perceived cognitive skills, the score calculation is evaluated as 0-none, 4-too much. Perceived cognitive disorders and perceived cognitive skills subsections contain opposite questions and the last 2 questions are not included in the scoring. The increase in the total score indicates the goodness of the situation in terms of cognitive functions.(Hospital group, telerehabilitation group and control group will be evaluated)
Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire | A day before the treatment
  The Arm, Shoulder and Hand Injuries Questionnaire (DASH) will be used to evaluate the functions of the upper extremities.This questionnaire assesses disability, activity limitations, restriction on leisure activities and participation in work. The DASH questionnaire consists of three parts. The first part consists of 30 questions. 21 questions determine the patient's difficulty during activities of daily living, five questions determine the symptoms (pain, activity-related pain, tingling, stiffness, weakness), each of the remaining four questions determine the social function, work, sleep and the patient's function /symptom score.(Hospital group, telerehabilitation group and control group will be evaluated)

SECONDARY OUTCOMES:
Chronic Disease Treatment Functional Assessment Fatigue (FACIT Fatigue) Scale | Baseline, 6 weeks, 12 weeks, and 6 months
  It is a measurement tool that subjectively evaluates the fatigue in the last week and consists of 13 expressions. The scale has a five-point Likert scale of 0 = not at all, 1 = very little, 2 = a little, 3 = a lot, and 4 = a lot. 11 items (1-6, 9-13) of the scale contain reverse expressions. The 7th and 8th items of the scale are calculated flat. The scores that can be obtained from the scale range from 0 to 52. A high total score on the scale indicates that the severity of fatigue is low. It is reported that the perception fatigue is clinically severe if the score from the scale is 30 or less. (Hospital group, telerehabilitation group and control group will be evaluated)
EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire) | 6 weeks, 12 weeks, and 6 months
  The EORTC-QLQ-C30 Quality of Life Scale includes 30 questions and three subheadings: general well-being, functional difficulties, and symptom control. The first 28 of the 30 items in the scale are a four-point Likert-type scale and the items are evaluated as Never: 1, A little: 2, Quite: 3 or A lot: 4 points. In the 29th question of the scale, the patient is asked to evaluate his health on a scale from 1 to 7 (1: Very poor and 7: Excellent), and in the 30th question, the general quality of life. The 29th and 30th questions constitute the general well-being area. High scores in this section indicate a high quality of life, and low scores indicate a decrease in quality of life. (Hospital group, telerehabilitation group and control group will be evaluated)
Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) | 6 weeks, 12 weeks, and 6 months
  This form evaluates the parameters of cognitive sensitivity (sharpness), attention and coordination, memory, verbal fluency, functional confusion, observations of others about the individual, change in functionality compared to before, and quality of life. It consists of 4 subtitles and 37 questions in total. Questions in the sections of perceived cognitive impairment, comments from other people, perceived cognitive skills, and impact on quality of life are scored between 0 and 4 (0-several times per day times, 4-never). In 9 questions in the field of perceived cognitive skills, the score calculation is evaluated as 0-none, 4-too much. Perceived cognitive disorders and perceived cognitive skills subsections contain opposite questions and the last 2 questions are not included in the scoring. The increase in the total score indicates the goodness of the situation in terms of cognitive functions.(Hospital group, telerehabilitation group and control group will be evaluated)
Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire | 6 weeks, 12 weeks, and 6 months
  The Arm, Shoulder and Hand Injuries Questionnaire (DASH) will be used to evaluate the functions of the upper extremities.This questionnaire assesses disability, activity limitations, restriction on leisure activities and participation in work. The DASH questionnaire consists of three parts. The first part consists of 30 questions. 21 questions determine the patient's difficulty during activities of daily living, five questions determine the symptoms (pain, activity-related pain, tingling, stiffness, weakness), each of the remaining four questions determine the social function, work, sleep and the patient's function /symptom score.(Hospital group, telerehabilitation group and control group will be evaluated)

CONTACTS AND LOCATIONS:
Locations (1):
- Ramazan Cihad Yılmaz, Gaziantep, Turkey (Türkiye)